CLINICAL TRIAL: NCT02076646
Title: A Phase I/II Dose Escalation Study of the Tumor-targeting Human L19-IL2 Monoclonal Antibody-cytokine Fusion Protein in Combination With Dacarbazine for Patients With Metastatic Melanoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19IL2DTIC-04-12
Record Dates: First submitted 2014-02-24; First posted 2014-03-03 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Melanoma Stage IV
Keywords: Interleukin; IL2; monoclonal; antibody; cytokine; Dacarbazine; metastatic; melanoma; tumor targeting; Dose definition; L19
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ph I: L19IL2 + DTIC (Experimental): Cohorts of 3-6 patients will receive escalating doses of L19-IL2 until MTD is reached.
  L19-IL2 will be administered on days 1, 8 & 15 of each 21-day-cycle. Dacarbazine will be given at a fixed dose on day 1 of each 21-day cycle, 30 minutes after the end of the L19-IL2 infusion.
  Interventions: Drug: L19IL2 - Ph I; Drug: DTIC
- Ph II - ARM 1: L19IL2 at RD + DTIC (Experimental): During the phase II part of this study, 60 patients with Stage IV M1a and M1b melanoma will be randomized in a 1:1 ratio: 30 patients assigned to Arm 1 will receive L19IL2 at the RD + DTIC at a fixed dose.
  Interventions: Drug: L19IL2 at RD - Ph II; Drug: DTIC
- Ph II - ARM 2: DTIC monotherapy (Active Comparator): During the phase II part of this study, 60 patients with Stage IV M1a and M1b melanoma will be randomized in a 1:1 ratio: 30 patients assigned to Arm 2 will receive DTIC at a fixed dose as monotherapy.
  Interventions: Drug: DTIC

INTERVENTIONS:
Drug: L19IL2 - Ph I — During phase I part of the study, increasing dose of L19IL2 from one cohort to the next will be performed in steps of 160,000 IU/kg starting at 480,000 IU/kg (i.e., 0.48; 0.64; 0.80 MioIU/kg until MTD is reached).
  Arms: Ph I: L19IL2 + DTIC
Drug: L19IL2 at RD - Ph II — L19IL2 at RD will be administered to Arm 1 patients during phase II part of the study.
  Arms: Ph II - ARM 1: L19IL2 at RD + DTIC
Drug: DTIC — Dacarbazine: 1 hour intravenous infusion on day 1 of each 21-cycle at a dosage of 1000 mg/m2 (fixed dose).
  Other Names: DETICENE®

SUMMARY:
A prospective, open-label, multi-center, Phase I/II study of L19IL2 in combination with Dacarbazine in patients with metastatic melanoma.

DETAILED DESCRIPTION:
A prospective, open-label, multi-center, Phase I/II dose escalation study in which cohorts of 3-6 patients with metastatic melanoma will be assigned to receive escalating doses of L19-IL2 in combination with a fixed dose of Dacarbazine.

After definition of MTD and RD during the phase II part of this study, 60 patients with Stage IV M1a and M1b melanoma will be randomized in a 1:1 ratio to receive open label the combination treatment at the RD (Arm 1) or DTIC monotherapy (Arm 2).

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years of age, inclusive
2. Must have histologically or cytologically confirmed cutaneous metastatic melanoma (Stage IV). For the Phase II part only patients with Stage IV M1a or M1b will be enrolled.
3. Must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) as identified by CT or MRI scan within 28 days before the first study drug administration.
4. Baseline LDH within normal range
5. Maximal 1 line of previous systemic treatment for metastatic disease (prior adjuvant melanoma therapy, e.g., IFN, is permitted.
6. For women of childbearing potential, a negative pregnancy test within 72 hours prior to the first dose of study treatment.
7. Women with reproductive potential must be willing to practice acceptable methods of birth control during the study and for up to 12 weeks after the last dose of study medication.
8. Men with reproductive potential must be willing to practice acceptable methods of birth control during the study and for up to 12 weeks after the last dose of study medication.
9. Must have Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
10. Life expectancy of at least three months
11. Adequate organ function: serum creatinine ≤ 1.5 x ULN, total bilirubin ≤ 30 mM/L (or mg/dL, ≤ 2.0 mg/dL), hepatic transaminases ≤ 2.5 x ULN, alkaline phosphatase ≤ 2.5 x ULN.
12. ANC count ≥ 1.5 x 10^9/L, platelet count ≥ 100 x 10^9/L, hemoglobin > 9 g/dL
13. Normal 12-lead ECG and normal bidimensional echocardiogram or MUGA
14. All toxic effects of prior therapy must have resolved to grade ≤1 unless otherwise specified above
15. Willing and able to give written informed consent.

Exclusion Criteria:

1. Pregnant or breastfeeding female
2. Primary ocular melanoma
3. Primary mucosal melanoma
4. Use of any investigational or other anti-cancer drug within 28 days or 5 half-lives, whichever is longer, preceding the first dose of DTIC and L19-IL2
5. Prior radiation to a target lesion, unless there has been clear progression of the lesion since radiotherapy
6. A history of known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection
7. History or clinical evidence of brain metastases or leptomeningeal disease
8. Any other malignancy from which the patient has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix
9. Treatment with DTIC within 6 months before start of study
10. Treatment with Ipilimumab within 6 months before start of study
11. Hypersensitivity to DTIC
12. Concomitant use of drugs known to alter cardiac conduction
13. Chronic use of corticosteroids used in the management of cancer or non-cancer-related illness
14. Unstable or serious concurrent uncontrolled medical conditions
15. Inadequately controlled cardiac arrhythmias including atrial fibrillation
16. History of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris
17. Heart insufficiency > grade II NYHA criteria
18. Uncontrolled hypertension
19. Ischemic peripheral vascular disease
20. Active infection or incomplete wound healing.
21. History or evidence of active autoimmune disease.
22. Known history of allergy to intravenously administered proteins/peptides/antibodies
23. History of organ allograft.or allogeneic peripheral blood progenitor cell or bone marrow transplantation
24. Major trauma including surgery within 4 weeks prior to entering the study.
25. Any underlying medical or psychiatric condition which in the opinion of the investigator will make administration of study drug hazardous or hinder the interpretation of study results (e.g. AE).
26. Melanoma patients with BRAF 600 E mutation who are amenable to receive approved treatments able to extend overall survival.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2013-07-31 (Actual); Primary Completion 2016-05-17 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Phase I: maximum tolerated dose (MTD) and recommended dose (RD) of L19IL2 | From day 1 to day 21 of Cycle 1 (each cycle is 21-days)
  Establish the MTD and the RD of L19IL2 (in combination with dacarbazine) to be used for phase II study
Phase II: best objective response rate (BORR) | Up to 1 year
  Evaluation of antitumor activity

SECONDARY OUTCOMES:
Phase I: best objective response rate (BORR) | Up to 1 year
  Evaluation of antitumor activity
Phase I: duration of objective response | From week 6 up to 1 year
  Evaluation of the antitumor activity
Phase I: disease control rate | At 6 months
  Evaluation of the antitumor activity
Phase I: median progression free survival (mPFS) | Up to 1 year
  Evaluation of the antitumor activity
Phase I: median overall survival and overall survival rate | Up to 1 year
  Evaluation of the antitumor activity
Phase II: safety and tolerability of L19-IL2 in combination with DTIC vs DTIC alone. | Up to 1 year
  Safety evaluation including AEs, SAE and standard laboratory assessment
Phase II: duration of objective response | Up to 1 year
Phase II: disease control rate | At 6 months
Phase II: median progression free survival (mPFS) | Up to 1 year
Phase II: median overall survival and overall survival rate | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Claus Garbe, Prof. M.D., Principal Investigator — University Hospital Tuebingen (Germany); Michele Maio, Dr.med., Principal Investigator — Azienda Ospedaliera Universitaria Senese, Siena (Italy)
Locations (2):
- University Hospital, Tübingen, Germany
- Azienda Ospedaliera Universitaria Senese, Siena, Italy